CLINICAL TRIAL: NCT07067307
Title: Clinical Evaluation of Melatonin Concomitant Use With Neoadjuvant Chemotherapy Protocols in Breast Cancer Patients
Brief Title: Melatonin in Breast Cancer Patients Receiving Neoadjuvant Chemotherapy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mona Mohammed El-Tamalawy, Lecturer of Clinical Pharmacy, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-104
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: melatonion; chemotherapy induced toxicity
MeSH Terms: conditions — Breast Neoplasms | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Active Comparator): Melatonin 20 mg once daily at bedtime
  Interventions: Drug: melatonin
- Control (Placebo Comparator): Placebo once daily at bedtime
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: melatonin — melatonin 20 mg tablet once daily at bedtime
  Arms: Melatonin
Drug: Placebo — Placebo once daily at bedtime
  Arms: Control

SUMMARY:
Melatonin is an attractive candidate with anticancer activities previously reported in various preclinical and clinical studies. Melatonin not only involves regulating biological rhythms and endocrine function but also functions in the occurrence, development, and treatment of cancer. There is a number of possible mechanisms by which melatonin may exert its anticancer effects. These mechanisms may include potent antioxidant, immunomodulating, oncostatic, antiproliferative, and estrogen-modulating properties. Regarding the immune-potentiating effects, melatonin increases the activity of lymphocytes, monocyte/ macrophage, and natural killer cells. Melatonin may also exert antiangiogenic and direct apoptotic effects. These activities, except for free-radical scavenging, are believed to be receptor-mediated through Melatonin-1 and Melatonin-2 receptors.

Preclinical studies have demonstrated the antitumor effects of melatonin when used alone and enhanced effects for chemotherapy when used in combination. Melatonin has shown positive results in a number of clinical trials on patients with cancer. The effect of melatonin in early stages and locally advanced breast cancer is still questioned.

Also the effect of melatonin on the development and severity of various chemotherapy-induced toxicities in breast cancer patients will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis with primary invasive breast cancer.
2. Patients eligible for receiving neoadjuvant chemotherapy.
3. Eastern Cooperative Oncology Group (ECOG) performance status from 0 to 2.
4. Adequate bone marrow function (white blood count ≥4,000/mm3, platelet count≥100,000/mm3), liver function (aspartate aminotransferase and alanine aminotransferase ≤ 2.5times the upper limit of normal, serum total bilirubin < 1.5 mg/dl), renal function (creatinine < 1.5 mg/dl)

Exclusion Criteria:

1. Patients with metastatic or non-invasive disease.
2. Patients previously received chemotherapy within one month preceding randomization.
3. Patients who were previously taking melatonin.
4. Hypersensitivity to melatonin.
5. Patients with autoimmune diseases.
6. Pregnancy and lactation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Response type to chemotherapy using Residual Cancer Burden (RCB) index. | At time of surgery after termination of neoadjuvant chemotherapy protocol
  Residual Cancer Burden index (RCB) is a validated, continuous index combining primary tumor size, cellularity, and nodal metastasis either pathological complete response or presence of residual tumor ( minimal, moderate, or extensive).
  The primary outcome is the difference in the mean or median RCB index between intervention and control group.

SECONDARY OUTCOMES:
Presence and density of Tumor Infiltrating Lymphocytes within the tumor tissue. | At time of surgery after termination of neoadjuvant chemotherapy protocol
  Difference between study arms regarding presence and density of Tumor Infiltrating Lymphocytes within the tumor tissue. This will reflect tumor's biology and the immune response it elicits.
The change in radiological tumor size | At time of surgery after termination of neoadjuvant chemotherapy protocol
  The change in radiological tumor size (expressed as the largest diameter) compared between both groups.
  The tumor size will be obtained from standard bilateral mammography and ultrasound imaging of the breast.
Incidence and grading of myelosuppression, mucositis, and peripheral sensory neuropathy | throughout the period of neoadjuvant chemotherapy protocol (about 6 months)
  Incidence of development and grading of some chemotherapy-induced toxicities (myelosuppression, mucositis, and peripheral sensory neuropathy) will be assessed using National Cancer Institute - Common Terminology Criteria for Adverse Events version 5
The proportion of patients achieving pathologic complete response (RCB-0) after neoadjuvant therapy in each group. | At surgery after completion of neoadjuvant chemotherapy.
Difference in proportions across RCB categories. | At surgery after completion of neoadjuvant therapy
  Comparison of the distribution of RCB categories (0, I, II, III) between intervention and control group.
  0: No residual disease, 1: minimal residual disease, II: moderate residual disease, III: Severe residual disease.

OTHER OUTCOMES:
Adverse effects | throughout the period of neoadjuvant chemotherapy protocol (about 6 months)
  Any adverse/side effect will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided